CLINICAL TRIAL: NCT05816668
Title: Tranexamic Acid's Effects in Patients Undergoing Laparoscopic Radical Prostatectomy: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Tranexamic Acid's Effects in Patients Undergoing Laparoscopic Radical Prostatectomy
Acronym: Transamin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, CAIO BRAMBILLA, MD, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NP2011/2021
Record Dates: First submitted 2022-12-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; video laparoscopic prostatectomy; tranexamic acid
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Just ICESP's Clinical Research Pharmacy team will be not blinded. The surgical and anesthetic teams will be blinded in relation to the placebo or tranexamic acid intervention during the preoperative period and during the postoperative follow-up and, if any case loses the blinding, it will be excluded from the analysis. The preparation of packaging, dilution and dispensing or the material containing tranexamic acid or placebo will be carried out by the ICESP's Clinical Research Pharmacy division.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Group (Experimental): Patients will receive an attack solution of 1,0 g of tranexamic acid 20 minutes before the surgery beginning, followed by a maintence dose of 1,0 mg/kg/h in pump surgery infusion
  Interventions: Drug: Tranexamic acid
- Placebo Group (Placebo Comparator): Patients undergoinf to videolaparoscopic surgery will receive physcological saline as placebo under the same conditions of the tranexamic acid group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Patients with prostate cancer and radical video laparoscopy prostatectomy indication will receive 1,0g of Tranexamic Acid solution IV in bolus 20 minutes before of anesthetic induction, followed by a maintenance hose of 1,0mg/kg/h of surgery.
  Other Names: Transamin
  Arms: Tranexamic Acid Group
Other: Placebo — Patients randomized to placebo group will receive physiological saline and will undergo to the radical video laparoscopu prostatectomy normally
  Arms: Placebo Group

SUMMARY:
The study is randomized, placebo-controlled, double-blind clinical trial that aims to check whether tranexamic acid's use in videolaparoscopic radical prostatectomy intraoperative is effective in decrease serum hemoglobin drop and the amount of blood's transfusion.

DETAILED DESCRIPTION:
The study aims to check whether tranexamic acid's use in videolaparoscopic radical prostatectomy intraoperative is effective in decrease serum hemoglobin drop and the amount of blood's transfusion.

Therefore it will be a randomized, placebo-controlled, double-blind clinical trial that intends to recruit 122 patients with radical prostatectomy indication who agreed to consent study inclusion.

Patients randomized to intervention group will receive 1,0g of tranexamic acid IV during anesthetic induction, followed by a maintenance dose of 1,0 mg/kg/hour of surgery. Control group will be operated normally.

Data as hemoglobin drop, estimated bleeding volume, need to transfusion, side effects, and presence of lymphocele will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years olds;
* Who accept to participate and sign the consent form;
* Compliance with the study follow-up protocol;
* Diagnosed with localized prostate cancer with surgical indication without or with lymphadenectomy.

Exclusion Criteria:

* Coronary artery disease treated with drug-using stent;
* Previous coronary procedures or coronary disease using a stent;
* Acute or chronic liver failure;
* Severe chronic renal failure (ClCr < 30 mL/Kg.h, according to the Modification of Diet in Renal Disease formula);
* Suspected allergy to tranexamic acid;
* Known coagulopathies and refusal to sign consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients diagnosed with localized prostate cancer
Enrollment: 122 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in serum Hemoglobin levels from preoperative to post operative levels | Baseline (Before) and 12 and 24 hours after surgery
  The serum hemoglobin drop will be evaluated

SECONDARY OUTCOMES:
Estimated volume of bleeding | During surgery
  Total blood loss will be assessed by the volume aspirated during surgery.
Transfusion rate of red blood cell concentrates | 12 and 24 hours after surgery
  The amount of red blood cells concentrate transfused will be evaluated.
Adverse effects tranexamic acid | Up to 30 days after surgery
  The adverse effects tranexamic acid administration will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ferreira Coelho, MD, PhD, Principal Investigator — Instituto do Câncer do Estado de São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Etzioni R, Tsodikov A, Mariotto A, Szabo A, Falcon S, Wegelin J, DiTommaso D, Karnofski K, Gulati R, Penson DF, Feuer E. Quantifying the role of PSA screening in the US prostate cancer mortality decline. Cancer Causes Control. 2008 Mar;19(2):175-81. doi: 10.1007/s10552-007-9083-8. Epub 2007 Nov 20. PMID 18027095
- [Background] Tsodikov A, Gulati R, Heijnsdijk EAM, Pinsky PF, Moss SM, Qiu S, de Carvalho TM, Hugosson J, Berg CD, Auvinen A, Andriole GL, Roobol MJ, Crawford ED, Nelen V, Kwiatkowski M, Zappa M, Lujan M, Villers A, Feuer EJ, de Koning HJ, Mariotto AB, Etzioni R. Reconciling the Effects of Screening on Prostate Cancer Mortality in the ERSPC and PLCO Trials. Ann Intern Med. 2017 Oct 3;167(7):449-455. doi: 10.7326/M16-2586. Epub 2017 Sep 5. PMID 28869989
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Cote K, Loffredo M, Schultz D, Chen MH, Tomaszewski JE, Renshaw AA, Wein A, Richie JP. Biochemical outcome after radical prostatectomy or external beam radiation therapy for patients with clinically localized prostate carcinoma in the prostate specific antigen era. Cancer. 2002 Jul 15;95(2):281-6. doi: 10.1002/cncr.10657. PMID 12124827
- [Background] Bekelman JE, Rumble RB, Chen RC, Pisansky TM, Finelli A, Feifer A, Nguyen PL, Loblaw DA, Tagawa ST, Gillessen S, Morgan TM, Liu G, Vapiwala N, Haluschak JJ, Stephenson A, Touijer K, Kungel T, Freedland SJ. Clinically Localized Prostate Cancer: ASCO Clinical Practice Guideline Endorsement of an American Urological Association/American Society for Radiation Oncology/Society of Urologic Oncology Guideline. J Clin Oncol. 2018 Nov 10;36(32):3251-3258. doi: 10.1200/JCO.18.00606. Epub 2018 Sep 5. PMID 30183466
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Rainwater LM, Segura JW. Technical consideration in radical retropubic prostatectomy: blood loss after ligation of dorsal venous complex. J Urol. 1990 Jun;143(6):1163-5. doi: 10.1016/s0022-5347(17)40215-1. PMID 2342176
- [Background] Ramsay C, Pickard R, Robertson C, Close A, Vale L, Armstrong N, Barocas DA, Eden CG, Fraser C, Gurung T, Jenkinson D, Jia X, Lam TB, Mowatt G, Neal DE, Robinson MC, Royle J, Rushton SP, Sharma P, Shirley MD, Soomro N. Systematic review and economic modelling of the relative clinical benefit and cost-effectiveness of laparoscopic surgery and robotic surgery for removal of the prostate in men with localised prostate cancer. Health Technol Assess. 2012;16(41):1-313. doi: 10.3310/hta16410. PMID 23127367
- [Background] Basiri A, de la Rosette JJ, Tabatabaei S, Woo HH, Laguna MP, Shemshaki H. Comparison of retropubic, laparoscopic and robotic radical prostatectomy: who is the winner? World J Urol. 2018 Apr;36(4):609-621. doi: 10.1007/s00345-018-2174-1. Epub 2018 Jan 23. PMID 29362896
- [Background] Rassweiler J, Hruza M, Teber D, Su LM. Laparoscopic and robotic assisted radical prostatectomy--critical analysis of the results. Eur Urol. 2006 Apr;49(4):612-24. doi: 10.1016/j.eururo.2005.12.054. Epub 2006 Jan 18. PMID 16442210
- [Background] Ilic D, Evans SM, Allan CA, Jung JH, Murphy D, Frydenberg M. Laparoscopic and robotic-assisted versus open radical prostatectomy for the treatment of localised prostate cancer. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD009625. doi: 10.1002/14651858.CD009625.pub2. PMID 28895658
- [Background] Mohler JL, Antonarakis ES, Armstrong AJ, D'Amico AV, Davis BJ, Dorff T, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Ippolito JE, Kane CJ, Kuettel MR, Lang JM, McKenney J, Netto G, Penson DF, Plimack ER, Pow-Sang JM, Pugh TJ, Richey S, Roach M, Rosenfeld S, Schaeffer E, Shabsigh A, Small EJ, Spratt DE, Srinivas S, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 May 1;17(5):479-505. doi: 10.6004/jnccn.2019.0023. PMID 31085757
- [Background] Tewari A, Srivasatava A, Menon M; Members of the VIP Team. A prospective comparison of radical retropubic and robot-assisted prostatectomy: experience in one institution. BJU Int. 2003 Aug;92(3):205-10. doi: 10.1046/j.1464-410x.2003.04311.x. PMID 12887468
- [Background] Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol. 2009 May;55(5):1037-63. doi: 10.1016/j.eururo.2009.01.036. Epub 2009 Jan 25. PMID 19185977
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Napolitano LM, Cohen MJ, Cotton BA, Schreiber MA, Moore EE. Tranexamic acid in trauma: how should we use it? J Trauma Acute Care Surg. 2013 Jun;74(6):1575-86. doi: 10.1097/TA.0b013e318292cc54. No abstract available. PMID 23694890
- [Background] Lin ZX, Woolf SK. Safety, Efficacy, and Cost-effectiveness of Tranexamic Acid in Orthopedic Surgery. Orthopedics. 2016 Mar-Apr;39(2):119-30. doi: 10.3928/01477447-20160301-05. Epub 2016 Mar 4. PMID 26942474
- [Background] Claeys MA, Vermeersch N, Haentjens P. Reduction of blood loss with tranexamic acid in primary total hip replacement surgery. Acta Chir Belg. 2007 Jul-Aug;107(4):397-401. doi: 10.1080/00015458.2007.11680081. PMID 17966532
- [Background] Dietrich W, Spannagl M, Boehm J, Hauner K, Braun S, Schuster T, Busley R. Tranexamic acid and aprotinin in primary cardiac operations: an analysis of 220 cardiac surgical patients treated with tranexamic acid or aprotinin. Anesth Analg. 2008 Nov;107(5):1469-78. doi: 10.1213/ane.0b013e318182252b. PMID 18931201
- [Background] MACFARLANE RG. AN ENZYME CASCADE IN THE BLOOD CLOTTING MECHANISM, AND ITS FUNCTION AS A BIOCHEMICAL AMPLIFIER. Nature. 1964 May 2;202:498-9. doi: 10.1038/202498a0. No abstract available. PMID 14167839
- [Background] DAVIE EW, RATNOFF OD. WATERFALL SEQUENCE FOR INTRINSIC BLOOD CLOTTING. Science. 1964 Sep 18;145(3638):1310-2. doi: 10.1126/science.145.3638.1310. PMID 14173416
- [Background] Wang YL, Jiang B, Yin FF, Shi HQ, Xu XD, Zheng SS, Wu S, Hou SC. Perioperative Blood Transfusion Promotes Worse Outcomes of Bladder Cancer after Radical Cystectomy: A Systematic Review and Meta-Analysis. PLoS One. 2015 Jun 16;10(6):e0130122. doi: 10.1371/journal.pone.0130122. eCollection 2015. PMID 26080092
- [Background] Linder BJ, Frank I, Cheville JC, Tollefson MK, Thompson RH, Tarrell RF, Thapa P, Boorjian SA. The impact of perioperative blood transfusion on cancer recurrence and survival following radical cystectomy. Eur Urol. 2013 May;63(5):839-45. doi: 10.1016/j.eururo.2013.01.004. Epub 2013 Jan 11. PMID 23332883
- [Background] Kerkebe Lama M, Orellana Salinas NR, Flores Martinez JM, Olivares Gribbell RA, Storme Cabrera O, Fuentealba Sudy CA. [Prospective study and comparative of surgical and oncologic outcome between laparoscopic and retropubical radical prostatectomy]. Actas Urol Esp. 2009 Feb;33(2):167-71. doi: 10.1016/s0210-4806(09)74118-x. Spanish. PMID 19418841
- [Background] Drouin SJ, Vaessen C, Hupertan V, Comperat E, Misrai V, Haertig A, Bitker MO, Chartier-Kastler E, Richard F, Roupret M. Comparison of mid-term carcinologic control obtained after open, laparoscopic, and robot-assisted radical prostatectomy for localized prostate cancer. World J Urol. 2009 Oct;27(5):599-605. doi: 10.1007/s00345-009-0379-z. Epub 2009 May 7. PMID 19421755
- [Background] Ficarra V, Novara G, Fracalanza S, D'Elia C, Secco S, Iafrate M, Cavalleri S, Artibani W. A prospective, non-randomized trial comparing robot-assisted laparoscopic and retropubic radical prostatectomy in one European institution. BJU Int. 2009 Aug;104(4):534-9. doi: 10.1111/j.1464-410X.2009.08419.x. Epub 2009 Mar 5. PMID 19281468
- [Background] Remzi M, Klingler HC, Tinzl MV, Fong YK, Lodde M, Kiss B, Marberger M. Morbidity of laparoscopic extraperitoneal versus transperitoneal radical prostatectomy verus open retropubic radical prostatectomy. Eur Urol. 2005 Jul;48(1):83-9; discussion 89. doi: 10.1016/j.eururo.2005.03.026. Epub 2005 Apr 12. PMID 15967256
- [Background] Ou YC, Yang CR, Wang J, Cheng CL, Patel VR. Comparison of robotic-assisted versus retropubic radical prostatectomy performed by a single surgeon. Anticancer Res. 2009 May;29(5):1637-42. PMID 19443379
- [Background] Batagello CA, Vicentini FC, Monga M, Miller AW, Marchini GS, Torricelli FCM, Danilovic A, Coelho RF, Srougi M, Nahas WC, Mazzucchi E. Tranexamic acid in patients with complex stones undergoing percutaneous nephrolithotomy: a randomised, double-blinded, placebo-controlled trial. BJU Int. 2022 Jan;129(1):35-47. doi: 10.1111/bju.15378. Epub 2021 Jun 13. PMID 33630393
- [Background] Crescenti A, Borghi G, Bignami E, Bertarelli G, Landoni G, Casiraghi GM, Briganti A, Montorsi F, Rigatti P, Zangrillo A. Intraoperative use of tranexamic acid to reduce transfusion rate in patients undergoing radical retropubic prostatectomy: double blind, randomised, placebo controlled trial. BMJ. 2011 Oct 19;343:d5701. doi: 10.1136/bmj.d5701. PMID 22012809
- [Background] Balik M, Kosina J, Husek P, Brodak M, Cecka F. Safety and Efficacy of Using Tranexamic Acid at the Beginning of Robotic-Assisted Radical Prostatectomy in a Double-Blind Prospective Randomized Pilot Study. Acta Medica (Hradec Kralove). 2020;63(4):176-182. doi: 10.14712/18059694.2020.60. PMID 33355078
- [Background] Saravanan R, Venkatraman R, Karthik K, Pushparani A. [Efficacy of different doses and timing of tranexamic acid in major orthopedic surgeries: a randomized trial]. Braz J Anesthesiol. 2020 Jul-Aug;70(4):311-317. doi: 10.1016/j.bjan.2020.03.013. Epub 2020 Jul 8. PMID 32753113
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912